CLINICAL TRIAL: NCT06734442
Title: Surgical Management of Primary Spontaneous Pneumothorax in Children
Brief Title: Thoracoscopy for Idiopathic Pneumothorax in Children
Acronym: THOPED
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Destinval Christelle, Dr., University Hospital, Clermont-Ferrand
Other Study IDs: M24DC1106; NCT05861037 (obsolete NCT alias)
Record Dates: First submitted 2024-12-11; First posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Spontaneous Pneumothorax; Idiopathic Pneumothorax; Bleb Lung; Child, Only
Keywords: Video-Assisted Thoracoscopy; Spontaneous Idiopathic Pneumothorax; Blebectomy; Lung Wedge; Pleural Abrasion; Retrospective Study; Child
MeSH Terms: conditions — Pneumothorax; Blister | interventions — Thoracic Surgery, Video-Assisted

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Video-Assisted Thoracoscopy with blebectomy and pleural abrasion — Thoracoscopic management of pneumothorax

SUMMARY:
The goal of this retrospective study is to describe the outcomes of spontaneous idiopathic pneumothorax treated by thoracoscopy with pleural abrasion and blebectomy.

The main questions it aims to answer are:

* are there risk factors leading to pneumothorax recurrence?
* are pleural abrasion and blebectomy really diminishing the recurrence of pneumothorax?

DETAILED DESCRIPTION:
The investigators describe the outcomes of the participants: length of stay, operating time, type and time before recurrence, occurrence of contralateral pneumothorax also treated by thoracoscopy, with pleural abrasion and blebectomy

ELIGIBILITY:
Inclusion Criteria:

* Patients younger than 18 years old who had a video-assisted thoracoscopy with pleural abrasion and blebectomy for spontaneous idiopathic pneumothorax

Exclusion Criteria:

* Patients older than 18 years old who had a video-assisted thoracoscopy with pleural abrasion and blebectomy for spontaneous idiopathic pneumothorax

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients who were operated from 2014 to 2022
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Recurrence of pneumothorax | Through study completion, an average of 2 years
  1. Recurrence of pneumothorax Recurrence of pneumothorax after first pleural drainage or persistant air leaking

SECONDARY OUTCOMES:
Other complications after surgery | Through study completion, an average of 2 years
  Hemothorax, early and late recurrence
Operating Time | Intraoperative
  Time for surgery
Length of stay | From admission to discharge home, up to 20 days
  Length of stay
The time between the surgery and postoperative consultation dates | Through study completion, an average of 2 years
  Follow-up represents the time between the surgery and postoperative consultation dates in days, months, or years.
  Generally, there are a-month-follow-up, a three month-follow-up, a six month-follow-up, and a year-follow-up. The surgeon can see the patient if there is any problem between these consultations. After a year of follow-up, it is up to the surgeon to decide if the patient needs to be seen yearly or not. The last follow-up date is crucial because it indicates how the patient is and if other follow-up dates need to be applied.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Clermont-Ferrand, Clermont-Ferrand, Auvergne, France

IPD SHARING:
Plan to Share IPD: No
In the name of anonymization the investigators won't share individual participant data

REFERENCES:
- [Background] Demir M, Akin M, Kaba M, Filiz S, Sever N, Karadag CA, Dokucu AI. Thoracoscopic Resection in the Treatment of Spontaneous Pneumothorax. Sisli Etfal Hastan Tip Bul. 2020 Mar 25;54(1):94-97. doi: 10.14744/SEMB.2018.88310. eCollection 2020. PMID 32377141
- [Background] Pogorelic Z, Gudelj R, Bjelanovic D, Jukic M, Elezovic Baloevic S, Glumac S, Furlan D. Management of the Pediatric Spontaneous Pneumothorax: The Role of Video-Assisted Thoracoscopic Surgery. J Laparoendosc Adv Surg Tech A. 2020 May;30(5):569-575. doi: 10.1089/lap.2019.0742. Epub 2020 Mar 11. PMID 32167851